CLINICAL TRIAL: NCT06273722
Title: Dynamic Optical Coherence Tomography for Detection and Subtyping of Basal Cell
Brief Title: D-OCT for Detection and Subtyping of BCC: a Diagnostic Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0059
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Basal Cell Carcinoma; Optical Coherence Tomography
Keywords: Basal cell carcinoma; Optical coherence tomography; Imaging; Non-melanoma skin cancer
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- D-OCT scanned patients: This diagnostic cohort study will include patients (18+ years) who underwent a biopsy and D-OCT scan for lesions suspect for BCC skin cancer. Patient data was retrieved from a pre-existing registry (METC: 2022-3555). All D-OCT scans were obtained at the outpatient dermatology clinic of Maastricht University Medical Center+ (MUMC+) using a Vivosight Multi-beam Swept-Source Frequency Domain OCT scanner (Michelson Diagnostics Maidstone, Kent, UK; resolution <7.5 µm lateral, <5 µm axial; depth of focus 1.0 mm; scan area 6 × 6 mm). All scanned lesions were histopathologically examined by a dermatopathologist blinded to D-OCT scans and D-OCT assessment.
  Interventions: Device: Vivosight Multi-beam Swept-Source Frequency Domain OCT scanner

INTERVENTIONS:
Device: Vivosight Multi-beam Swept-Source Frequency Domain OCT scanner — Vivosight Multi-beam Swept-Source Frequency Domain OCT scanner (Michelson Diagnostics Maidstone, Kent, UK; resolution <7.5 µm lateral, <5 µm axial; depth of focus 1.0 mm; scan area 6 × 6 mm).

SUMMARY:
The current gold standard for diagnosing basal cell carcinoma (BCC) is the histopathological examination of biopsy specimen. However, non-invasive imaging modalities such as optical coherence tomography (OCT) may replace biopsy if BCC presence and its subtype can be established with high confidence. Subtype differentiation is crucial; while superficial BCCs (sBCC) can be treated topically, nodular (nBCC) and infiltrative BCCs (iBCC) require excision. Dynamic OCT (D-OCT) is a functionality integrated within the OCT device, enabling the visualization of vascular structures through speckle variance.

Descriptive studies have unveiled vascular shapes and patterns associated with BCC and its respective subtypes. These findings suggest that D-OCT could contribute to the accuracy of BCC detection and subtyping. Yet comparative clinical studies between OCT and D-OCT are lacking. In the proposed diagnostic cohort study, we aim to assess whether D-OCT assessment is superior to OCT in terms of accuracy for BCC detection and subtyping.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years
* Lesions suspect for non-melanoma skin cancer or premalignancy
* Patient underwent D-OCT scan and biopsy conform regular care

Exclusion Criteria:

* Patient unable to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This diagnostic cohort study will include patients (18+ years) who underwent a biopsy and D-OCT scan for lesions suspect for BCC skin cancer. Patient data was retrieved from a pre-existing registry (METC: 2022-3555). All D-OCT scans were obtained at the outpatient dermatology clinic of Maastricht University Medical Center+ (MUMC+) using a Vivosight Multi-beam Swept-Source Frequency Domain OCT scanner (Michelson Diagnostics Maidstone, Kent, UK; resolution <7.5 µm lateral, <5 µm axial; depth of focus 1.0 mm; scan area 6 × 6 mm). All scanned lesions were histopathologically examined by a dermatopathologist blinded to D-OCT scans and D-OCT assessment.
Sampling Method: Non-Probability Sample
Enrollment: 424 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy for BCC detection on D-OCT assessment | Measured before December 31st 2024
  We will evaluate the ability of OCT assessors to discriminate BCC from non-BCC using OCT without and with dynamic functionality. The diagnostic certainty for BCC detection will be expressed on a five-point confidence scale. A high confidence score (confidence score=4) is considered a positive OCT test results. In these cases, biopsy could effectively be omitted. Lower confidence scores (confidence score≤3) are considered negative OCT test results as in these cases, biopsy remains necessary for a definitive or alternative diagnosis. The primary outcome of interest is the sensitivity of a high confidence BCC diagnosis because we want to evaluate whether the dynamic functionality increases the proportion of correctly classified BCCs.

SECONDARY OUTCOMES:
Diagnostic accuracy for BCC subtyping on D-OCT assessment | Measured before December 31st 2024
  We will evaluate the ability of OCT assessors to discriminate each individual BCC subtype from the other two subtypes using OCT without and with dynamic functionality. Cases that resulted in a high confidence diagnosis (confidence score=4) will be included in the analyses. Three analyses will be performed to calculate the sensitivity to detect sBCC, nBCC or iBCC and the specificity to identify non-sBCC, non-nBCC or non-iBCC subtypes using histopathology as reference test. In this respect, sensitivity is defined as the proportion of a specific BCC subtype, that is correctly classified as such by the OCT assessor (i.e. sBCC, nBCC or iBCC), whereas specificity is defined as the proportion of the other two subtypes that is correctly classified as such (i.e sBCC/nBCC, sBCC/iBCC or nBCC/iBCC). The primary outcome of interest is the sensitivity. We want to evaluate whether the dynamic functionality increases the proportion of correctly classified subtypes .
Diagnostic value of vascular structures and patterns | Measured before December 31st 2024
  Diagnostic odds ratios (DORs ) are used to identify subsets of vascular features and patterns that can be used to accurately discriminate BCC subtypes. The histopathological subtype (i.e. sBCC, nBCC, iBCC ) vs. other subtypes (i.e sBCC/nBCC, sBCC/iBCC, nBCC/iBCC) will be used as the dependent variable. A DOR >1 indicates that the presence of a vascular feature or pattern is indicative for the presence of the respective BCC subtype.

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared with other researchers upon reasonable request. Requests will be evaluated on a case by case manner.